CLINICAL TRIAL: NCT02558348
Title: A Phase 1/2a Evaluation of the Safety, Pharmacokinetics and Efficacy of AL3818, a Dual Receptor Tyrosine Kinase Inhibitor, in Subjects With Recurrent or Metastatic Endometrial, Ovarian or Cervical Cancer (AL3818-US-001)
Brief Title: Phase 1/2a Evaluation of AL3818 in Subjects With Recurrent or Metastatic Endometrial, Ovarian or Cervical Cancer (AL3818-US-001)
Acronym: AL3818
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor termination
Sponsor: Advenchen Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL3818-US-001
Record Dates: First submitted 2014-09-26; First posted 2015-09-24 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Endometrial Cancer; Ovarian Cancer; Cervical Cancer
Keywords: Dual receptor Tyrosine Kinase Inhibitor; Anti-angiogenic therapy
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AL3818 (Experimental): Part 1 (Phase 1b): Cohort 1 will initiate at a dose of 12 mg/day of AL3818, for 21-Day cycles (14 days of AL3818 treatment followed by 7 days of rest). After three subjects have completed the first cycle of therapy without a DLT, additional cohorts may be enrolled sequentially. After the first cohort has completed one full cycle of therapy without a DLT, two additional cohorts will be sequentially enrolled at 16 mg/day and 20 mg/day doses of AL3818 for the same 21-day cycles.
  Part 2 (Phase 2a): Each subject will receive a dose of up to 20 mg AL3818 or a maximum of the MTD from Part 1 (Phase 1b) of this study for continuous 21-Day cycles of therapy (14 days of AL3818 treatment followed by 7 days of rest).
  Interventions: Drug: AL3818

INTERVENTIONS:
Drug: AL3818 — Administered orally
  Other Names: Anlotinib Hydrochloride

SUMMARY:
The purpose of Part 1 (Phase 1b) is to evaluate the general safety and tolerability of repeated 21-day cycles of AL3818 therapy, and to reevaluate the maximum tolerated dose (MTD).

The purpose of Part 2 (Phase 2a) is to evaluate the efficacy of repeated 21-day cycles of AL3818 therapy preliminary efficacy of AL3818 in subjects with recurrent or metastatic endometrial, ovarian or cervical cancer.

DETAILED DESCRIPTION:
This is a Phase 1b/2a study to evaluate the safety, pharmacokinetics and efficacy of 21-day cycles of AL3818 therapy. The study is divided into two parts. Part 1 (Phase 1b) will evaluate the dose limiting toxicity (DLT) and general safety during the first 21-day cycle of Al3818 therapy and to reevaluate the MTD. It will include a sequential evaluation of 3 subjects per cohort in a 3+3 design with up to 18 subjects in total. Cohort 1 will initiate at a dose of 12 mg/day of AL3818, for cycles of 14 days of treatment followed by 7 days of rest. After three subjects have completed the first cycle of therapy without a DLT, additional cohorts may be enrolled sequentially. All subjects will be allowed continuation of therapy with repeat cycles of 21-days if they are tolerating AL3818 and have stable disease or better. After the first cohort has completed one full cycle of therapy without a DLT, two additional cohorts will be sequentially enrolled at 16 mg/day and 20 mg/day doses of AL3818 for the same 21-day cycles.

Part 2 (Phase 2a) will evaluate the safety and preliminary efficacy of repeated 21-day cycles of AL3818. It will include up to 45 additional subjects with metastatic endometrial cancer, ovarian cancer refractory to platinum therapy or cervical cancer refractory to standard therapy. Each subject will receive a dose of up to 20 mg AL3818 or a maximum of the MTD from Part 1 (Phase 1b) of this study for continuous 21-Day cycles of therapy (14 days of AL3818 treatment followed by 7 days off).

All subjects in Part 1 and Part 2 of this study will be permitted to continue therapy with only safety monitoring and bimonthly assessments for progression, if AL3818 is well tolerated and the subject has stable disease or better.

ELIGIBILITY:
Inclusion Criteria:

For a subject to be eligible for this study, she must meet all of the following criteria:

1. Female subjects 18 years of age or older
2. Subjects may be enrolled with previous histologically proven diagnosis of the following:

   a. Endometrial Cancer: Patients must have recurrent or persistent endometrial carcinoma, which is refractory to curative therapy or established treatments.

   i. Histologic diagnosis will be reviewed by the treating institution ii. Patients with the following histologic epithelial cell types are eligible: Endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified, mucinous adenocarcinoma, squamous cell carcinoma, and transitional cell carcinoma.

   iii. Initial treatment may have included chemotherapy, chemotherapy and radiation therapy, and/or consolidation/maintenance therapy; antiangiogenic therapy (e.g. bevacizumab) as part of adjuvant therapy is allowed. Chemotherapy administered in conjunction with primary radiation as a radio-sensitizer will be counted as a systemic chemotherapy regimen.

   iv. Patients should have received no more than two prior cytotoxic or non-cytotoxic therapies for management of recurrent or persistent disease (excluding endocrine therapies which will not count in the number of regimens)

   b. Ovarian cancer: Patients must have recurrent or persistent ovarian, fallopian tube or primary peritoneal cancer, which is refractory to established treatments.

   i. Patients with the following histologic epithelial cell types are eligible: Endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified.

   ii. Patients must have received at least one prior platinum-based chemotherapeutic regimen for the management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound.

   iii. This initial therapy may have included high-dose therapy, consolidation, or extended therapy administered after surgical or non-surgical assessment.

   iv. Antiangiogenic therapy (e.g. bevacizumab) as part of adjuvant therapy is allowed.

   v. Patients should have received no more than two prior cytotoxic or non-cytotoxic therapies for management of recurrent or persistent disease

   c. Cervix cancer: Subjects diagnosed with histologically confirmed squamous cell carcinoma of the cervix.

   i. Patients must have received at least one prior platinum based chemotherapeutic regimen for the management of primary disease containing carboplatin, cisplatin or another organoplatinum compound. The initial therapy may have included high-dose therapy, consolidation or extended therapy administered after surgical or non-surgical assessment. Antiangiogenic therapy (e.g. bevacizumab) as part of adjuvant therapy is allowed. Chemotherapy administered in conjunction with primary radiation as a radio-sensitizer will be counted as a systemic chemotherapy regimen.

   ii. Patients should have received no more than two prior cytotoxic or non-cytotoxic standard therapies for management of recurrent or persistent disease.

   d. Other uterine cancers: Subjects diagnosed with other uterine cancers, such as Leiomyosarcoma, and have received no more than two prior cytotoxic or non-cytotoxic standard therapies for management of recurrent or persistent disease.
3. For Phase 2a only, all patients must express at least one FGFr 1, 2 or 3 amplification (or mutation) from archived tissue or new biopsy. For non-amplified patients, approval of the site coordinator or the sponsor is required prior to enrollment.
4. All patients must have measurable disease. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded). Each lesion must be ≥ 20mm when measured by conventional techniques, including palpation, plain x-ray, CT, and MRI, or ≥ 10mm when measured by spiral CT.
5. Life expectancy ≥ 3 months
6. Subject must be suitable for oral administration of study medication
7. Patients must have signed an approved informed consent and authorization permitting release of personal health information.
8. Patient must have adequate:

   1. Bone Marrow Function: Absolute neutrophil count (ANC) greater then or equal to 1,500/mm3, equivalent to Common Toxicity Criteria (CTC) grade 1. Platelets greater than or equal to 100,000/mm3
   2. Renal Function: Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN), CTC grade 1. Note: If creatinine is greater than 1.5 x ULN, creatinine clearance must be greater than >50 mL/min.
   3. Hepatic Function: Bilirubin less than or equal to 1.5 x ULN (CTC grade 1) or less than or equal to 3.0 x ULN for subjects with Gilbert Syndrome; AST and ALT less than or equal to 3.0 ×ULN.
   4. Coagulation profile: PT such that international normalized ratio (INR) is ≤ 1.55 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin or low molecular weight heparin) and a PTT < 1.2 times control.
9. ECOG performance status ≤ 2.
10. Subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of AL3818 until 4 weeks after discontinuing study drug.
11. Subjects of child-bearing potential must have a negative serum pregnancy test prior to study entry and cannot be lactating.
12. Ability and willingness to comply with the study protocol for the duration of the study and with follow-up procedures.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from participation in the study:

1. Subjects who have received prior treatment with an FGFr inhibitor or antagonist of FGFr. Prior anti-VEGF or anti-angiogenic therapy is allowed in the adjuvant treatment setting Prior anti-VEGF or anti-angiogenic therapy for the treatment of recurrent disease is not allowed.
2. Patients who have received prior antiangiogenic therapy, including bevacizumab, sorafenib, sunitinib, in the setting of advanced disease.
3. Patients with serious, non-healing wound, ulcer or bone fracture.
4. Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels.
5. Patient with history or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases or history of cerebrovascular accident (CVA, stroke) transient ischemic attack (TIA) or subarachnoid hemorrhage within 6 months of the first date of treatment on this study.
6. However, patients with metastatic CNS tumors may participate in this trial, if the patient is > 4 weeks from therapy completion (including radiation and/or surgery), is clinically stable at the time of study entry and is not receiving corticosteroid therapy.
7. Patients with proteinuria. Patients discovered to have a urine protein of 1+ on dipstick or ≥ 30 mg/dl at baseline should undergo a 24-hour urine collection, which must be an adequate collection and must demonstrate < 1000 mg protein/24 hr to allow participation in the study.
8. Patients with clinically significant cardiovascular disease; this includes: Uncontrolled hypertension; Myocardial infarction or unstable angina within 6 months prior to registration; New York Heart Association (NYHA) Grade II or greater congestive heart failure (Appendix F); Serious cardiac arrhythmia requiring medication; Grade II or greater peripheral vascular disease (Appendix F).
9. Patients who are pregnant or nursing. To date, no fetal studies of AL3818 in animals or humans have been performed. Therefore, AL3818 should not be administered to pregnant women. Subjects will be apprised of the large potential risk to a developing fetus. It is not known whether AL3818 is excreted in human milk. Because many drugs are excreted in human milk, AL3818 should not be administered to nursing women. Women of childbearing potential must agree to use contraceptive measures during study therapy and for at least 3 months after completion of AL3818 therapy. Because many drugs are excreted in human milk.
10. Patients with uncontrolled hypokalemia, hypomagnesaemia, and/or hypocalcaemia.
11. Hemoptysis within 3 months prior to first scheduled dose of AL3818.
12. Patients with acute or chronic liver disease, active hepatitis A or B with known cirrhosis or liver dysfunction.
13. Cytotoxic chemotherapy, immunotherapy, or radiotherapy within 4 weeks (6 weeks in cases of mitomycin C, nitrosourea, lomustine) prior to first scheduled dose of AL3818 or a major surgical procedure within 28 days or minor surgical procedure performed within 7 days prior to first scheduled dose of AL3818.
14. Concomitant treatment with strong inhibitors or inducers of CYP3A4, CYP2C9 and CYP2C19 who cannot be switched to other alternative medications (See Appendix E).
15. Known history of human immunodeficiency virus infection (HIV).
16. Subjects with active bacterial infections (other than uncomplicated urinary tract infection) and/or receiving systemic antibiotics.
17. Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy.
18. History of non-malignant GI bleeding, gastric stress ulcerations, or peptic ulcer disease within the past 3-months that in the opinion of the investigator may place the patient at risk of side effects on an anti-angiogenesis product.
19. History of significant vascular disease (e.g. aortic aneurysm, aortic dissection).
20. Intra-abdominal abscess within the last 3 months.
21. History of uncontrolled hypertension that is not well managed by medication, as documented by 2 baseline evaluations taken one hour apart with systolic blood pressure >160 mm or diastolic blood pressure >90 mm Hg pressure, or that in the opinion of the investigator may place the patient at risk when taking a VEGF inhibitor.
22. Pre-existing uncontrolled hypertension as documented by 2 baseline BP readings taken at least one hour apart, defined as systolic bloodpressure (BP) >160 mm Hg or diastolic BP > 90 mm Hg pressure.
23. QTcF>470 msec on screening ECG.
24. A history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
25. The use of concomitant medications that prolong the QT/QTc interval.
26. Baseline echocardiogram (within 2 months) with left ventricular ejection fraction (LVEF) < 50%.
27. History of difficulty swallowing, malabsorption, active partial or complete bowel obstruction, or other chronic gastrointestinal disease or condition that may hamper compliance and/or absorption of AL3818.
28. History of pancreatitis and/or renal disease that includes histologically confirmed glomerulonephritis, biopsy proven tubulointerstitial nephritis, crystal nephropathy, or other renal insufficiencies.
29. Treatment with an investigational agent within the longest time frame of either 5 half- lives or 30 days of initiating study drug.
30. Known recreational substance abuse.
31. Known hypersensitivity to anti-angiogenic agents.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02-14 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability of 21-Day cycles of AL3818 measured by incidence and severity of treatment-related adverse events (TRAE) - Part 1 (Phase 1b) | Cycle 1 (21 Days)
  Incidence and severity of treatment-related adverse events reported and their relationship to AL3818 will be assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.3). Safety data will be tabulated and summarized and descriptive statistics will be provided for changes in vital signs, weight, clinical laboratory tests (serum chemistry and hematology) and electrocardiogram (ECG) results.
Maximum Tolerated Dose (MTD) - Part 1 (Phase 1b) | Cycle 1 (21 Days)
  Reevaluation of the MTD determined by DLT events
Objective Response Rates (ORR) - Part 2 (Phase 2a) | After every three complete 21-Day cycles of therapy (Day 64)
  Evaluation by Response Evaluation Criteria In Solid Tumors (RECIST, v1.1) criteria

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of plasma AL3818 - Part 1 (Phase 1b) | Cycle 1 only: Day 1 (30mins, 60mins, 2 hours, 4 hours and 24 hours [prior to dosing on Day 2] ), Day 15 and Day 22 (Prior to dosing)
  Maximum Plasma Concentration (Cmax)
Pharmacokinetics (PK) of plasma AL3818 - Part 1 (Phase 1b) | Cycle 1 only: Day 1 (30mins, 60mins, 2 hours, 4 hours and 24 hours [prior to dosing on Day 2] ), Day 15 and Day 22 (Prior to dosing)
  Area Under the Curve (AUC)
Clinical Benefit Rate (CBR) - Part 2 (Phase 2a) | After three 21-day cycles of treatment (Day 64)
  Evaluated by Response Evaluation Criteria In Solid Tumors (RECIST, v1.1) criteria after three complete 21-day cycles. Measured as CR+PR+SD (SD ≥ 16 weeks from inclusion)
Overall Survival (OS) - Part 2 (Phase 2a) | From the date the study treatment was initiated to the date of death, followed for 5 years.
  Overall survival is defined as the date the study treatment was initiated to the date of death from any cause. Kaplan-Meier analysis
Progression-Free Survival (PFS) rate - Part 2 (Phase 2a) | Duration of time from the start of treatment to the time of documented disease progression or death, whichever comes first, followed for 12 months.
  Evaluated by Response Evaluation Criteria In Solid Tumors (RECIST, v1.1) criteria after three complete 21-day cycles for up to 12 months. Kaplan-Meier analysis

OTHER OUTCOMES:
Determine fibroblast growth factor receptor (FGFr 1, 2 and 3) amplification (or mutation) status of each subject - Part 2 (Phase 2a) | Measured within 28 days of dosing on Day 1
  For participation in Phase 2a: FGFr amplification (or mutation) status of each subject will be determined by analyses of archived tissue or new biopsy (if archived tissue is unavailable) and correlate with response

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Advenchen Laboratories, LLC
Locations (2):
- United States (2):
  - University of Chicago Medical Center, Chicago, Illinois
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Niu G, Chen X. Vascular endothelial growth factor as an anti-angiogenic target for cancer therapy. Curr Drug Targets. 2010 Aug;11(8):1000-17. doi: 10.2174/138945010791591395. PMID 20426765
- [Background] Roskoski R Jr. Vascular endothelial growth factor (VEGF) signaling in tumor progression. Crit Rev Oncol Hematol. 2007 Jun;62(3):179-213. doi: 10.1016/j.critrevonc.2007.01.006. Epub 2007 Feb 26. PMID 17324579
- [Background] Dickson C, Spencer-Dene B, Dillon C, Fantl V. Tyrosine kinase signalling in breast cancer: fibroblast growth factors and their receptors. Breast Cancer Res. 2000;2(3):191-6. doi: 10.1186/bcr53. Epub 2000 Mar 25. PMID 11250709
- [Background] Cole C, Lau S, Backen A, Clamp A, Rushton G, Dive C, Hodgkinson C, McVey R, Kitchener H, Jayson GC. Inhibition of FGFR2 and FGFR1 increases cisplatin sensitivity in ovarian cancer. Cancer Biol Ther. 2010 Sep 1;10(5):495-504. doi: 10.4161/cbt.10.5.12585. Epub 2010 Sep 4. PMID 20595807
- [Background] Hoeben A, Landuyt B, Highley MS, Wildiers H, Van Oosterom AT, De Bruijn EA. Vascular endothelial growth factor and angiogenesis. Pharmacol Rev. 2004 Dec;56(4):549-80. doi: 10.1124/pr.56.4.3. PMID 15602010
- [Background] Kondo Y, Arii S, Mori A, Furutani M, Chiba T, Imamura M. Enhancement of angiogenesis, tumor growth, and metastasis by transfection of vascular endothelial growth factor into LoVo human colon cancer cell line. Clin Cancer Res. 2000 Feb;6(2):622-30. PMID 10690548
- [Background] Yeramian A, Moreno-Bueno G, Dolcet X, Catasus L, Abal M, Colas E, Reventos J, Palacios J, Prat J, Matias-Guiu X. Endometrial carcinoma: molecular alterations involved in tumor development and progression. Oncogene. 2013 Jan 24;32(4):403-13. doi: 10.1038/onc.2012.76. Epub 2012 Mar 19. PMID 22430211
- [Background] Byron SA, Loch DC, Pollock PM. Fibroblast growth factor receptor inhibition synergizes with Paclitaxel and Doxorubicin in endometrial cancer cells. Int J Gynecol Cancer. 2012 Nov;22(9):1517-26. doi: 10.1097/IGC.0b013e31826f6806. PMID 23060048
- [Background] Gorringe KL, Jacobs S, Thompson ER, Sridhar A, Qiu W, Choong DY, Campbell IG. High-resolution single nucleotide polymorphism array analysis of epithelial ovarian cancer reveals numerous microdeletions and amplifications. Clin Cancer Res. 2007 Aug 15;13(16):4731-9. doi: 10.1158/1078-0432.CCR-07-0502. PMID 17699850
- [Background] Christensen C, Lauridsen JB, Berezin V, Bock E, Kiselyov VV. The neural cell adhesion molecule binds to fibroblast growth factor receptor 2. FEBS Lett. 2006 Jun 12;580(14):3386-90. doi: 10.1016/j.febslet.2006.05.008. Epub 2006 May 11. PMID 16709412
- [Background] Byron SA, Gartside MG, Wellens CL, Goodfellow PJ, Birrer MJ, Campbell IG, Pollock PM. FGFR2 mutations are rare across histologic subtypes of ovarian cancer. Gynecol Oncol. 2010 Apr;117(1):125-9. doi: 10.1016/j.ygyno.2009.12.002. Epub 2010 Jan 27. PMID 20106510
- [Background] Taniguchi F, Itamochi H, Harada T, Terakawa N. Fibroblast growth factor receptor 2 expression may be involved in transformation of ovarian endometrioma to clear cell carcinoma of the ovary. Int J Gynecol Cancer. 2013 Jun;23(5):791-6. doi: 10.1097/IGC.0b013e31828f38c4. PMID 23640291
- [Background] Tsang TY, Mohapatral G, Itamochi H, Mok SC, and Birrer MJ., Abstract 1528: Identification of FGFR3 as a potential therapeutic target gene for human clear cell ovarian cancer by global genomic analysis. Proceedings: AACR Annual Meeting 2014; April 5-9, 2014; San Diego, CA
- [Background] Kawase R, Ishiwata T, Matsuda Y, Onda M, Kudo M, Takeshita T, Naito Z. Expression of fibroblast growth factor receptor 2 IIIc in human uterine cervical intraepithelial neoplasia and cervical cancer. Int J Oncol. 2010 Feb;36(2):331-40. PMID 20043066